CLINICAL TRIAL: NCT02907190
Title: Glycemic and Insulinemic Impact of Selected Canadian Beans
Acronym: MED-beans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guelph Food Research Centre (Other Government)
Collaborators: Glycemic Index Laboratories, Inc (Industry); Ontario Bean Growers Association (Unknown)
Responsible Party: Principal Investigator, Dan Ramdath, Research Scientist, Guelph Food Research Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GIL-1625-lentil study
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Impaired Glucose Tolerance
Keywords: pulses; beans; blood glucose; insulin
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bean Type (Experimental): Beans (black; cranberry; great northern; navy; pinto; red) soaked overnight and boiled. 1/2 cup serving eaten by participants at study visit
  Interventions: Other: Bean Type
- Starchy Foods (Active Comparator): 1/2 cup serving of rice or paste or potato or corn will be eaten by participants on different study visit
  Interventions: Other: Starchy Foods

INTERVENTIONS:
Other: Bean Type — 1/2 cup of freshly boiled beans will be eaten by participants on separate study visits
  Arms: Bean Type
Other: Starchy Foods — 1/2 cup serving of one of 4 starchy foods will be eaten by participants on different study visit
  Arms: Starchy Foods

SUMMARY:
The objective of this study is to compare the glycemic and insulinemic response elicited by ½ cup servings of 6 beans to those elicited by ½ cup servings of mashed potato, macaroni, rice and corn.

DETAILED DESCRIPTION:
In order for a food to be able to claim a reduced glycemic response, it must be shown that a typical serving of the food elicits a significantly lower blood glucose responses compared to a serving of an appropriate control food. While many studies have examined the GI of beans, few studies have compared the glycemic impact of a typical serving of beans to a typical serving of other starchy foods. Therefore, there are insufficient data to allow for a claim that beans have a low glycemic response. In addition, in order to make a claim of a reduced glycemic response, regulatory agencies also require that the insulinemic response to a food is not disproportionately increased.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant females, 18-75 years of age, inclusive
* Body mass index (BMI) < 40 kg/m²
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial and to refrain from smoking for 12hr prior to each visit.
* Normal fasting serum glucose (<7.0mmol/L capillary corresponding to whole blood glucose <6.3mmol/L).
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Known history of AIDS, hepatitis, diabetes or a heart condition
* Subjects using medications or with any condition which might, in the opinion of Dr. Wolever, the Medical Director of GI Labs, either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Major trauma or surgical event within 3 months of screening.
* Unwillingness or inability to comply with the experimental procedures and to follow GI Labs safety guidelines.
* Known intolerance, sensitivity or allergy to any ingredients in the study products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Glycemic Response | 120 minutes
  post prandial blood glucose response

SECONDARY OUTCOMES:
Insulin Response | 120 minutes
  post prandial blood insulin response

CONTACTS AND LOCATIONS:
Overall Officials: Dan Ramdath, PhD, Principal Investigator — GI Laboratories Inc.
Locations (1):
- Glycemic Index Laboratories, Inc, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] EFSA 2011: European Food Safety Authority, Scientific Opinion on the substantiation of health claims related to resistant starch and reduction of post-prandial glycaemic responses (ID 681), "digestive health benefits" (ID 682) and "favours a normal colon metabolism" (ID 783) pursuant to Article 13(1) of Regulation (EC) No 1924/20061. EFSA Journal 9(4):2024.
- [Background] EFSA: European Food Safety Authority, Panel on Dietetic Products, Nutrition and Allergies (NDA). 2012. Scientific Opinion. Guidance on the scientific requirements for health claims related to appetite ratings, weight management and blood glucose concentrations. EFSA Journal 10(3): 2604-2614.
- [Background] Health Canada. Bureau of Nutritional Sciences, food directorate, health products and food branch. June 2013. Draft guidance document on food health claims related to the reduction in post-prandial glycaemic response.
- [Background] Wolever TM, Jenkins DJ. The use of the glycemic index in predicting the blood glucose response to mixed meals. Am J Clin Nutr. 1986 Jan;43(1):167-72. doi: 10.1093/ajcn/43.1.167. PMID 3942088
- [Background] Wolever TMS (2006). The Glycaemic Index: A Physiological Classification of Dietary Carbohydrate. CABI Publishing, Wallingford, UK.
- [Background] Ramdath D, Renwick S, Duncan AM. The Role of Pulses in the Dietary Management of Diabetes. Can J Diabetes. 2016 Aug;40(4):355-63. doi: 10.1016/j.jcjd.2016.05.015. PMID 27497151